CLINICAL TRIAL: NCT05166343
Title: Pediatric Out-of-Hospital Cardiac Arrest Resuscitation: Evaluation of IM Epinephrine (The PRIME Trial)
Brief Title: POHCA Resuscitation: Evaluation of IM Epinephrine
Acronym: PRIME
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Janice Tijssen, MD MSc, Interim Director, Paediatric Critical Care, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRIME-1
Record Dates: First submitted 2021-11-22; First posted 2021-12-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Out-of-Hospital Cardiac Arrest
Keywords: cardiac arrest; IM Epinephrine; standard of care; pediatric; resuscitation
MeSH Terms: conditions — Heart Arrest | interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: Paramedic services across Ontario will participate in the study. All sites will begin with a period of baseline data collection (standard of care arm) and will cross over to the intervention arm (Intramuscular Epinephrine Dose arm) on a staggered schedule and in random order. Each site will remain in the intervention arm, once cross over happens, for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): All POHCA events will be handled per standard of care of epinephrine administration via intravenous or intraosseous (IV/IO) based on patient estimated weight.
- Intramuscular Epinephrine Dose (Other): POHCA events will be handled per standard of care, however, first dose epinephrine administration will be via intramuscular (IM) autoinjector and/or pre-filled syringes. Dosing will be dependent on weight as follows:
  * 3-<5kg=0.3mg IM epinephrine
  * 5-<10kg=0.5mg IM epinephrine
  * 10-<20kg=1.0mg IM epinephrine
  * 20-<30kg=2.0mg IM epinephrine
  * 30kg=3.0mg IM epinephrine
  Interventions: Drug: Epinephrine Injection

INTERVENTIONS:
Drug: Epinephrine Injection — Epinephrine administered via sterile epinephrine injection USP, by 0.3mg or 0.5mg epinephrine auto-injector(s) and/or pre-filled syringe (exact dose).
  Arms: Intramuscular Epinephrine Dose

SUMMARY:
This is a pragmatic, two-arm, open-label, prospective stepped-wedge cluster quasi randomized control trial (SW-CRCT) looking to evaluate early intramuscular (IM) epinephrine in the management of pediatric out-of-hospital cardiac arrest (POHCA).

DETAILED DESCRIPTION:
IM epinephrine may provide a more efficient means of administering the initial epinephrine dose (versus IV/IO administration) to a child experiencing pediatric out of hospital cardiac arrest (POHCA) with no greater risk of harm. In so doing, this may improve the short- and long-term outcomes of these patients. There is an abundance of literature detailing the risk/benefit profile of IM epinephrine use in anaphylaxis; however, there is no human data on this topic as it relates to cardiac arrest. Important knowledge gaps include whether the use of IM epinephrine via autoinjector and/or pre-filled syringe leads to faster administration of the initial doses of epinephrine without delaying time to definitive epinephrine (via IV/IO) and the impact on time to initial and sustained return of spontaneous circulation (ROSC). This trial will be the first to examine the role of IM epinephrine via autoinjector/pre-filled syringe in POHCA.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 day to and including 17 years experiencing an out-of-hospital cardiac arrest (OHCA)
* Must be receiving at least 1 minute of CPR by trained first responders (police, fire, or paramedic services)

Exclusion Criteria:

- Children who experience OHCA due to an obvious traumatic event.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 284 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Time to initial return of spontaneous circulation (ROSC) | At time of event
  The primary outcome will be the time to initial ROSC. The investigator will compare time to initial ROSC between the standard of care and intervention periods.

SECONDARY OUTCOMES:
Return of spontaneous circulation | At time of event
  Whether return of spontaneous circulation is achieved or not
Time to sustained ROSC | At time of event
  Time to sustained ROSC will be calculated from the time that paramedics arrive on scene to the time that sustained ROSC, defined as chest compressions not required for 20 minutes with persistent signs of circulation, is achieved.
Survival | From time of event to ED admission
  Survival to emergency department transfer to pediatric critical care unit (PCCU), if applicable: admitted to PCCU from external ED
Survival - comparison between both arms | From time of event to hospital admission
  Survival to hospital admission will be compared between standard of care and intervention periods
PCCU/Hospital length of stay | From time of hospital/PCCU admission to discharge, up to 1 year
  PCCU and hospital length of stay will be calculated from time of admission to the PCCU/hospital and time to discharge from PCCU/hospital, if applicable, between standard of care and intervention periods
Survival to hospital discharge | Dependent on course of hospital stay, up to 1 year
  Survival to hospital discharge will be compared between standard of care and intervention periods
Post POHCA survival | Dependent on survival at 6 and 12 month period post POHCA event
  Survival at 6 months and 12 months post-POHCA will be compared between standard of care and intervention periods
Neurological status | From time of discharge and 6 and 12 months post POHCA event
  The investigator will compare PCPC scores at discharge, 6- and 12-months post-POHCA between the standard of care and intervention periods
Life Impact and Pediatric Quality of Life assessments | 6 and 12 months post POHCA event
  Life Impact assessment between 6 and 12 months: the investigator will use the Pediatric Quality of Life (PEDSQoL, Pediatrics Quality of Life) assessment tool at 6- and 12-months post-POHCA in all survivors and compare between standard of care and intervention periods. The score ranges from 0-100, with higher scores indicating better outcome.
Life Impact and Pediatric Quality of Life assessments | 6 and 12 months post POHCA event
  Life Impact assessment between 6 and 12 months: the investigator will use the Daily Activities Scale at 6- and 12-months post-POHCA in all survivors and compare between standard of care and intervention periods. This scale is a subscore of the PEDSQoL tool with scores ranging from 0-100, with higher scores indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tijssen, MD MSc, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Children's Hospital - London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No